CLINICAL TRIAL: NCT04325945
Title: Taipei Veterans General Hospital,Taiwan, R.O.C.
Brief Title: Evaluation of Laser Acupuncture on Health Promotion of Sub-health People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Director, Center for Traditional Medicine, Principal Investigator, Assistant Professor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-01-026CCF
Record Dates: First submitted 2020-03-18; First posted 2020-03-30 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Suboptimal Health Status
Keywords: pre-hypertension; insomnia; obesity
MeSH Terms: conditions — Prehypertension; Sleep Initiation and Maintenance Disorders; Obesity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture (Experimental): 808nm low level laser therapy
  Interventions: Device: Low level laser therapy
- Sham laser acupuncture (Sham Comparator): no low level laser output but same device
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Low level laser therapy — 808nm low level laser therapy on acupuncture points

SUMMARY:
Background: Suboptimal health status (SHS) is a dynamic state wherein people have not been diagnosed with a disease but tend to develop diseases. People with SHS often experience fatigue and other nonspecific symptoms. Early TCM-based interventions in people with SHS can prevent them from developing chronic diseases, thereby reducing the burden on health insurance systems. No study has explored the effects of laser acupuncture (LA) on people with SHS.

Material and Methods: Thirty SHS subjects with pre-hypertension or/and insomnia or/and obesity will be enrolled and assigned into a experiment group and a control group randomly in the first year protocol. One week before the start of the experiment, we will use questionnaires and mobile cloud-based devices to assess the physical status, such as blood pressure, body mass index, waist girth, hips girth, blood oxygen saturation, physical activity, pulse signal, autonomic nervous function, and sleep patterns. The subjects in the treatment groups received LA and those in control group received sham LA for 15 minutes per session twice a week for 8 weeks (16 sessions totally). All questionnaires, physical status and objective sleep parameters will be assessed in treatment group and control group after the 16th session. In the second year protocol, seventy SHS subjects will be enrolled and same procedure will be performed as the first year protocol.

DETAILED DESCRIPTION:
Background: Suboptimal health status (SHS) is a dynamic state. The term refers to an existing condition of ill health that could lead to a pathological condition but could also be eliminated, enabling the individual in question to return to a state of good health.

Traditional Chinese medicine (TCM) emphasizes the importance of health care and the idea that preventive treatment for diseases is superior to curative treatment. Therefore, TCM intervention will be eliminated SHS becoming to a chronic disease. According to previous studies, people with SHS without sports habits have 8 times risk of developing hypertension. In addition, people with SHS have more rates of sleep disorders, which are associated with obstructive sleep apnea due to decreased oxygen maturation during sleep, than healthy subjects.

A cloud TCM health-care model, which is combined with constitution patterns in TCM and physiological parameters, applied to Taiwanese with SHS. Taiwanese with SHS, no matter yang deficiency, Ying deficiency or Phlegm-stasis patterns, have decreased cardiac parasympathetic activity and high frequency change in pulse power spectrum analysis at right Chi. This phenomenon implied that people with SHS reduced convergence of the ministerial fire in the gate of life and then developed a disharmonic status between "Heart" and "Kidney" in TCM. This theory can explain why SHS has sleep disorders and prehypertension.

Laser acupuncture (LA) has been used in preventive diseases and many effects. Modern researches showed LA improved insomnia, circulation, analgesia and metabolism. However, it is still lacking evidences of objective parameters of sleep and there are no studies about TCM patterns change in SHS by LA.

In this study, the effects of 8 weeks' LA intervention on people with SHS presented with pre-hypertension and/or sleep disorders by a cloud health-care system combined with TCM patterns and physiological parameters will be investigated by 2-years protocols. The result will be helpful to establish the role of LA for preventive medicine in Taiwan.

Hypothesis: Regular LA intervention can improve sleep quality and regulate blood pressure and autonomic nervous function of sub-healthy people. Moreover, combining the cloud-based TCM body constitution and physical healthcare system can help sub-healthy people manage their own health better.

Material and Methods: Thirty SHS subjects with pre-hypertension or/and insomnia or/and obesity will be enrolled and will be assigned into a experiment group and a control group randomly in the first year protocol. One week before the start of the experiment, we will use questionnaires and mobile cloud-based devices to assess the physical status, such as blood pressure, body mass index, waist girth, hips girth, blood oxygen saturation, physical activity, pulse signal, autonomic nervous function, and sleep patterns. The subjects in the treatment groups received LA and those in control group received sham LA for 15 minutes per session twice a week for 8 weeks (16 sessions totally). All questionnaires will assessed in treatment group and control group before the first session and after the 16th session. In addition, we using mobile cloud-based devices to assess the physical status, such as blood pressure, blood oxygen saturation, physical activity, pulse signal, tongue examination, and autonomic nervous function before and after each sessions. Furthermore, sleep patterns will assessed for at least 2 days.

In the second year protocol, seventy SHS subjects with pre-hypertension or/and insomnia or/and obesity will be enrolled. and assigned into a experiment group and a control group randomly. The evaluation methods are the same as the first year protocol. Besides, we will build up the cloudy system to present body constitution scores and objective parameters. The auto-feedback function will be established in the second year protocol.

ELIGIBILITY:
Inclusion Criteria:

* Measure blood pressure at rest 120-139 / 80-89 mmHg more than 3 times a week.

PSQI score greater than 5.

Body mass index (BMI) :24~30 Kg/m2

Exclusion Criteria:

* Patients diagnosed with chronic diseases, such as hypertension, diabetes, chronic hepatitis, chronic kidney disease, chronic hyperlipidemia, coronary heart disease and other diseases that fall into the scope of chronic diseases of universal health insurance.

Diagnosis of mental illness.

Cancer patient

Pregnancy

People with significant inflammation at the time of participation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Change from Baseline Systolic Blood Pressure at 5 and 8 weeks
Body mass index | Change from Baseline Body Mass Index at 5 and 8 weeks
Sleep quality | Change from Baseline Sleep Quality Index at 5 and 8 weeks
  Pittsburgh sleep quality index

SECONDARY OUTCOMES:
Brain waves | Change from Baseline Brain Waves at 5 and 8 weeks
  Delta activity (0.5-4 Hz)、Theta activity (4-7 Hz) and alpha activity
Heart rate variability | Change from Baseline Heart Rate Variability at 5 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ying Kung, MD, Principal Investigator — Center for Traditional Medicine,Taipei Veterans General Hospital
Locations (1):
- Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei, Taiwan